CLINICAL TRIAL: NCT04816435
Title: Review of Classical Predictors and Role of Airway Ultrasound in the Prediction of Difficult Airway
Brief Title: Airway Ultrasound Assessment in the Prediction of Difficult Airway
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Other Study IDs: FJD-ECOVAD-01
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Airway Complication of Anesthesia; Anesthesia Intubation Complication
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound test — Ultrasound evaluation of airway

SUMMARY:
To assess whether the thickness of pre-tracheal fat, greater than 28 mm, and measured by ultrasound, constitutes a reliable parameter in the prediction of a difficult airway.

ELIGIBILITY:
Inclusion Criteria:

* Patients risk ASA I-IV
* Non-urgent surgery under general anesthesia with orotracheal intubation
* Acceptance to participate and grant written consent

Exclusion Criteria:

* Urgent surgery
* Patients with a history of craniocervical pathology (trauma, tumor, malformations)
* Pregnancy
* Patient Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients under general anesthesia with orotracheal intubation
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Pretracheal fat thickness for intubation complexity | 5 minutes
  The pretracheal fat at the level of the vocal cords will be evaluated with ultrasound, to discern if a certain thickness is related to a difficult laryngoscopic vision (understood as cormack 3 or 4)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Fundación Jimenez Díaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Madrid-Vazquez L, Casans-Frances R, Gomez-Rios MA, Cabrera-Sucre ML, Granacher PP, Munoz-Alameda LE. Machine learning models based on ultrasound and physical examination for airway assessment. Rev Esp Anestesiol Reanim (Engl Ed). 2024 Oct;71(8):563-569. doi: 10.1016/j.redare.2024.05.006. Epub 2024 May 31. PMID 38825182